CLINICAL TRIAL: NCT04659382
Title: A Prospective, Multicenter, Open-label, Phase II Study to Evaluate Efficacy and Safety of Selective Internal Radiation Therapy Plus Xelox, Bevacizumab and Atezolizumab (Immune Chekpoint Inhibitor) in Patients With Liver-dominant Metastatic Colorectal Cancer
Brief Title: Study to Evaluate Efficacy and Safety of Selective Internal Radiation Therapy Plus Xelox, Bevacizumab and Atezolizumab (Immune Chekpoint Inhibitor) in Patients With Liver-dominant Metastatic Colorectal Cancer
Acronym: SIRTCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD1709-SIRTCI
Record Dates: First submitted 2020-11-30; First posted 2020-12-09 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Colorectal Cancer; pMMR; MSS; Immune Checkpoint Inhibitor; Internal Radiotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — atezolizumab; XELOX; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): XELOX + bevacizumab + atezolizumab + SIRT (Therasphere)
  Interventions: Drug: Atezolizumab; Device: Therasphere; Drug: XELOX; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab combined to standard chemotherapy (XELOX + bevacizumab) and targeted therapy in patients whose tumour has been made immunogenic by radiotherapy (Therasphere) and ICI (atezolizumab).
Device: Therasphere — Therasphere injected to patients to promote the release of neoantigens from their tumour and convert it into an immunogenic tumour.
Drug: XELOX — standard chemotherapy for first line treament of metastatic CRC (in pMMR and/or MSS patients)
Drug: Bevacizumab — standard targeted therapy associated with XELOX for first line treament of metastatic CRC (in pMMR and/or MSS patients)

SUMMARY:
The main objective of the SIRTCI study is to evaluate the safety and efficacy of the combination chemotherapy (XELOX: Capecitabine plus oxaliplatin), anti-angiogenic (Bevacizumab), SIRT (TheraSphere®) and ICI (Atezolizumab) in patients with CRC with predominant liver metastases. SIRTCI is a single-arm, prospective, multi-centre phase II study. The main inclusion criteria are patients with MSS mRCC with predominantly non-operable liver metastases and measurable disease. Patients with extra-hepatic metastases can be included since the objective of the study is to induce local and abscopal effects of radiotherapy combined with ICI by stimulating the anti-tumour immune response to destroy both hepatic and extra-hepatic metastases.

DETAILED DESCRIPTION:
About 50% of patients with CRC will develop a metastatic disease. Majority of patients have unresectable disease and unresectable liver-dominant disease represents 25% of all mCRC. Morbidity and mortality in patients with mCRC are mainly due to unresectable liver metastases. In this setting, chemotherapy (doublet or triplet) plus biological agent remains the standard of care since no prospective randomized trial demonstrates the efficacy of local treatments (chemoembolization or hepatic arterial infusion chemotherapy). Actually median PFS in patients with unresectable liver-dominant mCRC is range between 9 to 12 months and more effective treatments must be evaluated.

ICI are to date ineffective in pMMR mCRC due to low level of tumor mutational load. Nevertheless, radiation induces an immunogenic cell death able to convert a "nonimmunogenic" neoplasm into an "immunogenic" neoplasm. In patients with liver-dominant mCRC SIRT has not shown survival improvement but only delayed disease progression in the liver. ICI improve efficacy of radiation both in irradiated lesions and non-irradiated lesions (abscopal effect). One explanation of the absence of PFS improvement with SIRT in first-line setting could be the progression of the extra-hepatic disease. Indeed, the rationale of SIRTCI 01 is to combine SIRT and ICI to induce an immune response and an abscopal effect against mCRC in order to improve control of hepatic disease (increase local SIRT efficacy with ICI) and extra-hepatic disease (increase abscopal effects of SIRT with ICI).

The aim of this study is therefore to demonstrate the synergistic anti-tumor efficacy of SIRT and ICI in patients with unresectable liver-dominant mCRC. Primary endpoint is PFS at 9 months. Main secondary endpoints are safety, response rate and OS. In addition, exploratory biomarker analyses will be performed in order to identify predictive factors of SIRT plus ICI efficacy. No safety issue was observed with XELOX/bevacizumab/atezolizumab and SIRT/FOLFOX/bevacizumab then the combination evaluated in SIRTCI 01 should be safe. Moreover oxaliplatin dose is decreased before SIRT treatment and bevacizumab is added only after SIRT treatment. All well-known predictive biomarkers of chemotherapy (mutational status, circulating tumor DNA) and ICI (tumor mutational load, immune response) efficacy will be analyzed. Additionally, pharmacokinetic analyses of Atezolizumab and centralized imaging review will be performed to evaluate morphologic and metabolic predictive markers (CT-scan, MRI, FDG PET/CT and Y90 PET/CT) of SIRT plus ICI efficacy.

This study will be the first one to use SIRT in order to induce immunogenic cell death and sensitivity to ICI. Combination of SIRT and ICI could increase immune abscopal anti-tumor effects of radiation. Indeed, once activated in one place (liver), the immune system can attack tumor lesions anywhere else in the body (lung, peritoneum…) through this abscopal effect.

SIRTCI 01 will provide informations on efficacy and safety of SIRT, ICI and chemotherapy combination in patients with unresectable liver-dominant mCRC. SIRT plus chemotherapy as well as chemotherapy plus ICI are well tolerated. TheraSphere® will be administered 3 or 4 days after cycle 2 or 3 of chemotherapy with adaptation of chemotherapy doses. Moreover, an interim analysis is planned to access efficacy of the strategy (first step after 22 evaluable patients included). At the time of the interim analysis, a complete review of the toxicities will be done to check the safety of the strategy and an independent data monitoring committee will monitor in real time all severe adverse events.

PFS at 9 months has been chosen as primary endpoint because it is a surrogate marker of OS. Actually median PFS in first-line setting with a doublet plus a biological agent is range from 8 to 11 months in unresectable mCRC and 9 to 12 months in unresectable liver-dominant mCRC, corresponding to a PFS of 50%-60% at 9 months. PFS is more reliable than response rate at 2-3 months given that the treatments used can induce tumor necrosis (SIRT) and/or initial pseudo-progression (ICI). In addition, most of patients will have a disease control/response at 2-3 months with this combination.As in all innovative phase II trials, this study should well include selected patients . A randomized phase II study with a large population does not seem appropriate in view of the limited literature on the safety and efficacy of this combination. The alternative clinical hypothesis to obtain 70% of patients alive and without progression at 9 months is ambitious and currently not achieved with current chemotherapies plus a biological agent.

The study will include patients with liver-dominant disease. Nevertheless, since the aim of the trial is to induce immune abscopal anti-tumor effects of radiation, patients with hepatic and extra-hepatic lesions will be included; extrahepatic lesions will be permitted if they are not symptomatic and if there is no organ dysfunction (up to 10 lesions). As ICI are very effective in dMMR mCRC (marketing authorization ongoing) it has been decided to exclude patients with dMMR mCRC.

The PFS obtain in SIRTCI 01 will provided a rationale for a randomized phase III study comparing chemotherapy alone (doublet or triplet ± biological agent) versus chemotherapy, SIRT and ICI combination in mCRC patients with unresectable liver-dominant disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically proven mismatch repair proficient metastatic colorectal cancer (pMMR and/or MSS)
* Liver-dominant disease with up to 6 extrahepatic lesions (only peritoneal lesions are not allowed) if asymptomatic and without organ dysfunction.
* Measurable disease according to RECIST 1.1
* Patient with initially unresectable disease according to the local multidisciplinary team and eligible for radioembolization according to the radiologist's opinion
* Tumor volume < 50 % of total liver volume
* No prior oncologic treatment for metastatic disease (i.e. chemotherapy, radiotherapy or investigational drug). Patients may have received adjuvant chemotherapy or (neo) adjuvant radiochemotherapy to the pelvis (tumor of the rectum), but the last dose of chemotherapy/radiotherapy must be administered at least 6 months prior to entry into this study. Analgesic radiotherapy of metastasis is permitted except on hepatic lesions and must be completed at least 14 days before inclusion.
* WHO performance status ≤ 1
* Estimated life expectancy ≥ 3 months
* Adequate hematological function: with neutrophils ≥ 1,500 /mm3, platelet count ≥ 100,000/mm3, hemoglobin > 9 g/dL (5,6 mmol/l)
* Adequate hepatic function: hepatic transaminases (ASAT and ALAT) ≤ 5 x UNL, total bilirubin ≤ 2 x UNL, alkaline phosphatase ≤ 5 x UNL
* Adequate renal function: creatinine clearance ≥ 50 ml/min according MDRD (Modification of Diet in Renal Disease)
* Patient affiliated to a social security system Information provided to patient and signature of the informed consent form by patient and the investigator

Exclusion Criteria:

* Active infection still requiring intravenous antibiotics on the first scheduled day of protocol treatment
* Symptomatic or untreated central nervous system metastasis
* Medical history of other concomitant or previous malignant disease, except adequately treated in situ carcinoma of the uterine cervix, basal or squamous cell carcinoma of the skin, or cancer in complete remission for ≥ 5 years,
* Other malignancy in the 5 years prior to inclusion in the study, except for localized cancer in situ, basal or squamous cell skin cancer
* Confirmed peritoneal carcinomatosis (lesions detectable on CT-scan and/or MRI)
* Active autoimmune disease or inflammatory bowel disease
* Bone marrow allograft or solid organ transplant history
* History of idiopathic pulmonary fibrosis, drug-induced pneumonitis or evidence of active pneumonitis on screening chest CT-scan and any severe chronic respiratory insufficiency that the investigator believes would not allow the SIRT to be received safely
* Positive tests for HIV or other immunodeficiency syndromes
* Severe chronic liver failure, which in the investigator's opinion would not allow SIRT to be received safely
* Active hepatitis B or hepatitis C.
* Active tuberculosis
* Patient with contraindication to angiography and selective hepatic catheterization such as bleeding diathesis or coagulopathy with serious bleeding risk that is not correctable by usual therapy of hemostatic agents.
* Patients on anticoagulant therapy different from low-molecular-weight heparin (LMWH) cannot be included (i.e. VKA and NOACs). Relaying these anticoagulants to a LMWH before inclusion is allowed. In addition, it must be possible to stop the LMWH 24 hours before invasive procedures according to the usual recommendations (before the work-up and before the SIRT).
* Significant presence of ascites, cirrhosis, portal hypertension, main portal venous tumor involvement or thrombosis on clinical or radiological evaluation Previous radiotherapy in the upper abdominal region (liver or liver vessels in the radiation field)
* If primary tumor is non-resected, it must be asymptomatic
* Long-term immunosuppressant therapy (patients requiring corticosteroid therapy are eligible if they receive a dose equivalent to no more than 10 mg of prednisone equivalent dose per day, and corticosteroid administration is permitted by a route resulting in minimal systemic exposure (cutaneous, rectal, articular, ocular or inhalation) is authorized)
* Partial or complete DPD deficiency
* Known hypersensitivity to any components of bevacizumab, Chinese Hamster Ovary cell products or other recombinant human or humanized antibodies and any other contraindications to the use of investigational medicinal products, in particular patients with peripheral sensory neuropathy with functional impairment (see SmPC of oxaliplatin) or in the case of recent or concomitant treatment with brivudine (see SmPC of capecitabine)
* QT/QTc interval > 450 msec for male and > 470 msec for female at EKC.
* K+ < LLN, Mg²+ < LLN, Ca²+ < LLN
* Allergy to contrast agents that do not allow radioembolization to be performed
* Uncontrolled hypertension (blood pressure > 140 mm Hg and/or diastolic blood pressure > 90 mm Hg)
* Clinically significant cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to the start of study treatment, myocardial infarction ≤ 6 months prior to the start of study treatment, unstable angina, congestive heart failure of NYHA (New York Heart Association Functional Classification) grade 2 or higher, or severe cardiac arrhythmia not controlled by drug therapy or which may interfere with study treatment
* Significant vascular disease (e.g. aortic aneurysm requiring surgery or arterial thrombosis) within 6 months prior to initiation of study treatment
* Venous thromboembolic disease within 3 months prior to initiation of study treatment
* Surgical procedure (including surgical biopsy, any surgical resection, or other major surgery) or significant traumatic injury within 28 days prior to start of study treatment, or planning major surgery during the study.
* History of abdominal fistula, gastrointestinal (GI) perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to start of study treatment
* Unhealing decaying wound, active ulcer, or untreated bone fracture
* Proteinuria ≥ 2+ by urine dipstick unless a 24-hour urine protein < 1 g of protein is demonstrated
* Lack of effective contraception in patients (male and/or female) at risk of reproduction, pregnant or breastfeeding women and women at risk of reproduction who have not had a pregnancy test.
* Persons deprived of freedom or under guardianship
* Inability to undergo medical follow-up of the study for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 9 months | 9 months after inclusion of the last patient
  The main objective of this study is to evaluate the progression-free survival at 9 months (according to RECIST 1.1) according to the investigator.

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - Chu - Hôpital Sud, Amiens
  - Privé - Cac - Clinique Bergonié, Bordeaux
  - Chu - Hôpital Henri Mondor, Créteil
  - Chu - Hôpital François Mitterrand, Dijon
  - Privé - Cac - Centre Georges François Leclerc, Dijon
  - Chu - Hôpital Grenoble Alpes, Grenoble
  - Chu - Hôpital Edouard Herriot, Lyon
  - Chu - Hôpital La Timone, Marseille
  - Privé - Cac - Institut Paoli Calmettes, Marseille
  - Chu - Hôpital Saint Éloi, Montpellier
  - Chu - Hôpital Européen Georges Pompidou, Paris
  - Chu - Hôpital Saint Louis, Paris
  - Chu - Hôpital Haut Lévêque, Pessac
  - Chu - Hôpital Lyon Sud, Pierre-Bénite
  - Chu - Hôpital La Milétrie, Poitiers
  - Privé - Cac - Centre Eugène Marquis, Rennes
  - Chu - Hôpital Charles Nicolle, Rouen
  - Privé - Cac - Centre Henri Becquerel, Rouen
  - Chu - Hôpital Hautepierre, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wasan HS, Gibbs P, Sharma NK, Taieb J, Heinemann V, Ricke J, Peeters M, Findlay M, Weaver A, Mills J, Wilson C, Adams R, Francis A, Moschandreas J, Virdee PS, Dutton P, Love S, Gebski V, Gray A; FOXFIRE trial investigators; SIRFLOX trial investigators; FOXFIRE-Global trial investigators; van Hazel G, Sharma RA. First-line selective internal radiotherapy plus chemotherapy versus chemotherapy alone in patients with liver metastases from colorectal cancer (FOXFIRE, SIRFLOX, and FOXFIRE-Global): a combined analysis of three multicentre, randomised, phase 3 trials. Lancet Oncol. 2017 Sep;18(9):1159-1171. doi: 10.1016/S1470-2045(17)30457-6. Epub 2017 Aug 3. PMID 28781171
- [Background] Venook AP, Niedzwiecki D, Lenz HJ, Innocenti F, Fruth B, Meyerhardt JA, Schrag D, Greene C, O'Neil BH, Atkins JN, Berry S, Polite BN, O'Reilly EM, Goldberg RM, Hochster HS, Schilsky RL, Bertagnolli MM, El-Khoueiry AB, Watson P, Benson AB 3rd, Mulkerin DL, Mayer RJ, Blanke C. Effect of First-Line Chemotherapy Combined With Cetuximab or Bevacizumab on Overall Survival in Patients With KRAS Wild-Type Advanced or Metastatic Colorectal Cancer: A Randomized Clinical Trial. JAMA. 2017 Jun 20;317(23):2392-2401. doi: 10.1001/jama.2017.7105. PMID 28632865
- [Background] Heinemann V, von Weikersthal LF, Decker T, Kiani A, Vehling-Kaiser U, Al-Batran SE, Heintges T, Lerchenmuller C, Kahl C, Seipelt G, Kullmann F, Stauch M, Scheithauer W, Hielscher J, Scholz M, Muller S, Link H, Niederle N, Rost A, Hoffkes HG, Moehler M, Lindig RU, Modest DP, Rossius L, Kirchner T, Jung A, Stintzing S. FOLFIRI plus cetuximab versus FOLFIRI plus bevacizumab as first-line treatment for patients with metastatic colorectal cancer (FIRE-3): a randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Sep;15(10):1065-75. doi: 10.1016/S1470-2045(14)70330-4. Epub 2014 Jul 31. PMID 25088940
- [Background] Saltz LB, Clarke S, Diaz-Rubio E, Scheithauer W, Figer A, Wong R, Koski S, Lichinitser M, Yang TS, Rivera F, Couture F, Sirzen F, Cassidy J. Bevacizumab in combination with oxaliplatin-based chemotherapy as first-line therapy in metastatic colorectal cancer: a randomized phase III study. J Clin Oncol. 2008 Apr 20;26(12):2013-9. doi: 10.1200/JCO.2007.14.9930. PMID 18421054
- [Background] Loupakis F, Cremolini C, Masi G, Lonardi S, Zagonel V, Salvatore L, Cortesi E, Tomasello G, Ronzoni M, Spadi R, Zaniboni A, Tonini G, Buonadonna A, Amoroso D, Chiara S, Carlomagno C, Boni C, Allegrini G, Boni L, Falcone A. Initial therapy with FOLFOXIRI and bevacizumab for metastatic colorectal cancer. N Engl J Med. 2014 Oct 23;371(17):1609-18. doi: 10.1056/NEJMoa1403108. PMID 25337750
- [Background] van Hazel GA, Heinemann V, Sharma NK, Findlay MP, Ricke J, Peeters M, Perez D, Robinson BA, Strickland AH, Ferguson T, Rodriguez J, Kroning H, Wolf I, Ganju V, Walpole E, Boucher E, Tichler T, Shacham-Shmueli E, Powell A, Eliadis P, Isaacs R, Price D, Moeslein F, Taieb J, Bower G, Gebski V, Van Buskirk M, Cade DN, Thurston K, Gibbs P. SIRFLOX: Randomized Phase III Trial Comparing First-Line mFOLFOX6 (Plus or Minus Bevacizumab) Versus mFOLFOX6 (Plus or Minus Bevacizumab) Plus Selective Internal Radiation Therapy in Patients With Metastatic Colorectal Cancer. J Clin Oncol. 2016 May 20;34(15):1723-31. doi: 10.1200/JCO.2015.66.1181. Epub 2016 Feb 22. PMID 26903575
- [Background] Gruenberger T, Bridgewater J, Chau I, Garcia Alfonso P, Rivoire M, Mudan S, Lasserre S, Hermann F, Waterkamp D, Adam R. Bevacizumab plus mFOLFOX-6 or FOLFOXIRI in patients with initially unresectable liver metastases from colorectal cancer: the OLIVIA multinational randomised phase II trial. Ann Oncol. 2015 Apr;26(4):702-708. doi: 10.1093/annonc/mdu580. Epub 2014 Dec 23. PMID 25538173